CLINICAL TRIAL: NCT04071964
Title: Gut Microbiota, Anastomotic Leak and Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 19.021-YP,2020-8305
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: Microbiota
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Groupe 1: Patients with colorectal cancer undergoing resection with anastomosis
- Groupe 2: Patients with colorectal cancer undergoing resection without anastomosis (Abdominoperineal resection)
- Groupe 3: Patients with rectal cancer without surgery ("Watch and wait")
- Groupe 4: Control group consisting of patients who do not have surgical pathologies of the colon and rectum

SUMMARY:
This is a prospective study evaluating the relation between the gut microbiota composition, intestinal healing after colorectal surgery and colorectal cancer behavior.

Our hypothesis is that the gut microbiota composition could predict poor intestinal healing in colorectal surgery, and that the gut microbiota might have an impact on colorectal cancer clinical behavior and may predict disease outcomes.

DETAILED DESCRIPTION:
No more details required

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* CRC diagnosis
* Upcoming colonic and/or rectal resection with/without anastomosis
* Individuals without diseases of the colon and rectum (healthy controls)

Exclusion Criteria:

* Pregnancy
* Previous stoma
* Bowel surgery in the last 4 weeks prior to the surgery

Secondary objectives, inclusion criteria are as follows:

* Age 18 years and older
* Rectal cancer diagnosis with histopathological confirmation
* Abdominoperineal resection with terminal colostomy
* Expectative non-surgical management ("Watch and wait approach")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer undergoing surgical resection (or expectative management for rectal cancer after complete clinical response to chemoradiotherapy)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2025-07-09 (Estimated); Study Completion 2025-07-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with an anastomotic leak | 1 month
  Clinical and/or radiological anastomotic leak

SECONDARY OUTCOMES:
Number of participants with cancer reoccurence | 3 years
  Colorectal cancer local or distant reoccurence

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada